CLINICAL TRIAL: NCT02724293
Title: Analgesic Efficacy and Safety of Peri-operative Pregabalin Following Radical Cystectomy, a Prospective,Randomized, Double-blinded, Controlled Trial
Brief Title: Efficacy and Safety of Peri-operative Pregabalin After Radical Cystectomy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmad Mohammad Abd El-Rahman, Lecturer of anesthesia, icu, and pain management, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 266
Record Dates: First submitted 2016-03-25; First posted 2016-03-31 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Postoperative Pain Following Radical Cystectomy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group I (placebo) (Placebo Comparator): patients received placebo.
  Interventions: Drug: placebo
- Group II (pregabaline 300 once) (Active Comparator): patients received pregabalin 300 mg 2 hours preoperatively.
  Interventions: Drug: pregabaline 300 mg once.
- Group III (pregabaline 300 twice) (Active Comparator): patients received pregabalin 300 mg 2 hours preoperatively and 12 hours after the preoperative dose.
  Interventions: Drug: pregabaline 300 mg twice.
- Group IV (pregabaline 600) (Active Comparator): patients received pregabalin 600 mg 2 hours preoperatively
  Interventions: Drug: pregabaline 600 mg once.

INTERVENTIONS:
Drug: pregabaline 300 mg once. — patients received pregabaline 300 mg 2 hours pre-operatively.
  Arms: Group II (pregabaline 300 once)
Drug: pregabaline 300 mg twice. — patients received pregabaline 300 mg 2 hours pre-operatively, and 12 hours later.
  Arms: Group III (pregabaline 300 twice)
Drug: pregabaline 600 mg once. — patients received pregabaline 600 mg 2 hours pre-operatively.
  Arms: Group IV (pregabaline 600)
Drug: placebo — patients received placebo
  Arms: Group I (placebo)

SUMMARY:
This study compares analgesic efficacy, and safety of three different doses of peri-operative pregabaline to placebo following radical cystectomy.

ELIGIBILITY:
Inclusion Criteria:

* Sixty patients between the ages of 18 and 60 years.
* American Society of Anesthesiologists (ASA) I-II physical status.
* undergoing radical cystectomy under general anesthesia.

Exclusion Criteria:

* Patients with a history of drug or alcohol abuse.
* patients with chronic pain or daily intake of analgesics.
* uncontrolled diabetes mellitus.
* uncontrolled hypertension.
* atherosclerotic heart disease.
* seizures.
* impaired kidney or liver functions,
* patients with body mass index ≥35 kg/m2, and whom
* patients that could not control a patient controlled analgesia (PCA) device.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2014-09; Primary Completion 2015-10 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
visual analogue scale (VAS) score | 24 hours postoperatively
  analgesic efficacy of study drugs as represented by the VAS score of the patients in the first 24 hours.
postoperative opioid consumption | 24 hours postoperatively
  ability of study drugs to reduce the postoperative opioid analgesic consumption.
time to first request of opioid analgesia | 24 hours postoperatively
  ability of the study drugs to delay the request of rescue opioid analgesia.

SECONDARY OUTCOMES:
Safety assessed by incidence of side effects | 24 hours postoperatively
  represented by the incidence of side effects during the follow up period of 24 hours.